CLINICAL TRIAL: NCT05341245
Title: Graphene Oxide in the Surgical Management of Intrabony Periodontal Defects: A Randomized Experimental Study With Histomorphometric Analysis
Brief Title: Graphene Oxide in the Surgical Management of Intrabony Periodontal Defects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Zeiad Khaled, Principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1091
Record Dates: First submitted 2022-03-22; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases | interventions — graphene oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Graphene oxide group (Experimental): The surgical defect will be managed by open flap debridement and application of Graphene oxide
  Interventions: Procedure: Graphene oxide and open flap debridement
- Open flap group (Other): The surgical defect will be managed by open flap debridement
  Interventions: Procedure: Open flap debridement

INTERVENTIONS:
Procedure: Graphene oxide and open flap debridement — Using Graphene oxide with open flap debridement in management of periodontal intrabony defects in dogs
  Arms: Graphene oxide group
Procedure: Open flap debridement — Using Open flap debridement in management of periodontal intrabony defects in dogs
  Arms: Open flap group

SUMMARY:
Using Graphene oxide in the surgical management of periodontal intrabony defects.

DETAILED DESCRIPTION:
Evaluation of the effect of Graphene oxide in the surgical management of periodontal intrabony defects in animals in periodontal clinical parameters with histomorphometric evaluation .

ELIGIBILITY:
Inclusion Criteria:

* male dogs
* 12-24 months old with approximate weight of 20-30 kg and general good health will be used

Exclusion Criteria:

-

Ages: 1 Year to 2 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
periodontal probing depth | 2 months
  To evaluate the use of Graphene Oxide in the surgical management of intrabony periodontal defects regarding the changes in periodontal probing depth "measured in mm " using University of North Carolina periodontal probe( UNC 15 probe ).
Clinical attachment level | 2 month
  To evaluate the use of Graphene Oxide in the surgical management of intrabony periodontal defects regarding the changes in clinical attachment level "measured in mm " using University of North Carolina periodontal probe( UNC 15 probe )

SECONDARY OUTCOMES:
Histomorphometric evaluation | 2 months
  To evaluate the use of Graphene Oxide in the surgical management of intrabony periodontal defects using histological sections obtained from the surgical site to do quantitative assessment of bone remodeling, modeling, and structure by "counting the number of osteoblasts and the number of bone trabeculae " using computer based microscope and software.

IPD SHARING:
Plan to Share IPD: Undecided